CLINICAL TRIAL: NCT00527865
Title: Study 181-1-06-01 - Phase 1A Clinical Study With DAS181: Double-Blind, Randomized, Placebo-Controlled, Single Dose Escalating Study in Healthy Adults
Brief Title: Single Dose Escalating Study of DAS181 in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Mang Yu, Nexbio, Inc
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-0082; 181-1-06-01; NCT00718900 (obsolete NCT alias)
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Influenza
Keywords: Influenza, Flu, DAS181, Fludase
MeSH Terms: conditions — Influenza, Human | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): 6 subjects DAS181 dosage 0.5 mg; 3 subjects placebo
  Interventions: Drug: DAS181; Drug: Placebo
- 2 (Experimental): 6 subjects DAS181 dosage 1.0 mg; 3 subjects placebo
  Interventions: Drug: DAS181; Drug: Placebo
- 3 (Experimental): 6 subjects DAS181 dosage 2.25 mg; 3 subjects placebo
  Interventions: Drug: DAS181; Drug: Placebo
- 4 (Experimental): 6 subjects DAS181 dosage 4.5 mg; 3 subjects placebo
  Interventions: Drug: DAS181; Drug: Placebo

INTERVENTIONS:
Drug: DAS181 — DAS181 is formulated as dry powder and packaged in capsules containing DAS181. The delivered dose of DAS181 dry powder at each fill size is 0.5 mg, 1.0 mg, 2.25 mg, and 4.5 mg.
Drug: Placebo — Capsules containing 10.5 mg of lactose will be supplied as placebo.

SUMMARY:
This study will evaluate the safety, tolerability, and systemic exposure of an experimental influenza (flu) treatment medication called DAS181. DAS181 is a dry powder that is administered via oral inhalation using a special device. Study participants will include up to 60 healthy, non-smoking males and females, ages 18-65. They will be given either DAS181 or placebo. Participants will remain in the clinic overnight to be watched for health changes for 24 hours after receiving the medication. Study procedures include: physical exams, chest x-rays, ECGs, lung function tests, collection of blood and urine samples, and throat swabs. Follow-up visits will occur on study days 2, 7, 14 +/- 1 day, and 30 +/- 2 days. Participants will be involved in the study for up to 61 days, which includes the screening period.

DETAILED DESCRIPTION:
The objective of this study is to investigate the safety, tolerability and pharmacokinetics of a single dose of DAS181 encapsulated dry powder compared to placebo when administered by oral inhalation using a dry powder inhaler in healthy adults. Primary study outcome measures are the safety and tolerability of single-dose DAS181 treatment at 0.5 mg, 1.0 mg, 2.25 mg, and 4.5 mg, as measured in the following parameters: adverse events, physical exam, vital signs, hematology, clinical chemistry, blood coagulation, complement activation, haptoglobin and immunogenicity, urinalysis, throat swab for bacterial culture, ECG, chest X-ray, and spirometric lung function. Secondary outcome measures are the systemic exposure and pharmacokinetic parameters of DAS181. This phase 1 study will be a double-blind, randomized, placebo-controlled, single-dose escalation study conducted at Comprehensive Phase One Miramar campus. Thirty-six to 60 healthy male and female volunteers, 18-65 years (inclusive), will be enrolled in 4 separate steps. Each enrollment will recruit 9 subjects for one of the 4 dose groups. Within each dose group, the participants will be randomly assigned to placebo or DAS181, at 1:2 ratios. The subjects will receive a single-dose treatment by placebo (10.5 mg lactose), or by DAS181 at one of 4 doses: 0.5 mg, 1.0 mg, 2.25 mg, and 4.5 mg. The subjects will be screened and enrolled within 28 days prior to dosing of the study drug. The study will be initiated with 0.5 mg dose. Escalation to the next dose will be contingent upon meeting the dose escalation criteria after the study day 7 post dosing follow-up visit (Visit 4). The day of dosing is always defined as Day 0 (or study day 0), regardless of the step or cohort. All future visits and time periods are referenced to the day of dosing. Administration of DAS181 or placebo will be given under the supervision of the study staff. Subjects will enter the inpatient clinic on day -1, the evening prior to dosing. Subjects will remain in the inpatient clinic for 24 hours post exposure to be observed for signs of adverse events (AEs). After the 24-hour inpatient observation period, participants will be discharged if they are deemed healthy at that point. All subjects must come back for follow-up visits on the following study days: 2, 7, 14 (±1 day), and 30 (±2 days).

ELIGIBILITY:
Healthy, non-smoking adult male and female volunteers between the ages of 18 and 65(inclusive)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single-dose of DAS181 treatment at 0.5 mg, 1.0 mg, 2.25 mg, and 4.5 mg. | Duration of study

SECONDARY OUTCOMES:
The pharmacokinetic parameters of DAS181. | Pre-dosing, 1, 2, 4, 6, 8, 12 and 24 hours post dosing, Day 2, and Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States

REFERENCES:
- [Derived] Zenilman JM, Fuchs EJ, Hendrix CW, Radebaugh C, Jurao R, Nayak SU, Hamilton RG, McLeod Griffiss J. Phase 1 clinical trials of DAS181, an inhaled sialidase, in healthy adults. Antiviral Res. 2015 Nov;123:114-9. doi: 10.1016/j.antiviral.2015.09.008. Epub 2015 Sep 25. PMID 26391974
- See also: NexBio, Inc — http://www.nexbio.com